CLINICAL TRIAL: NCT04850976
Title: Self-Assembled Modified Macintosh Videolaryngoscope Versus McGrath Macintosh (MAC®) Videolaryngoscope: Which is Better?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Raden Besthadi Sukmono, Anesthesiologist, Regional Anesthesia Consultant, Assistant Professor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IndonesiaUniv
Record Dates: First submitted 2021-04-08; First posted 2021-04-20 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Airway Management
Keywords: endotracheal intubation; self-assembled videolaryngoscope; McGrath MAC®; intubation time; glottis visualization
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Intervention Model Description: There were 2 intervention groups: (1) the Self-Assembled Modified Macintosh Videolaryngoscope (SAM-VL) group or (2) the McGrath MAC ® videolaryngoscope (McGrath) group.
Who Masked: Participant, Investigator
Masking Description: Randomization was done with tables and then presented in a closed envelope when the patient arrived at the operating room to determine the intervention group: (1) the Self-Assembled Modified Macintosh Videolaryngoscope (SAM-VL) group or (2) the McGrath MAC ® videolaryngoscope (McGrath) group. The laryngoscopist is the one who opened the envelope. A research assistant helped to prepare the laryngoscope according to the randomization results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Assembled Modified Macintosh Videolaryngoscope (SAM-VL) group (Experimental): The self-assembled modified Macintosh videolaryngoscope (SAM-VL) used in this study was constructed from a portable video camera with Wi-fi connection (Wi-fi Endoscope Video Camera model YPC99) attached to a no. 4 Macintosh Laryngoscope blade (Riester® no.7040). The video signal is transmitted to an Android-based mobile phone (Android version 7.0). The portable 2 megapixels video camera is 8 mm in diameter with 8 Light Emitting Diode (LED) lights for adjustable lighting level and 3 meters cable length. Video resolution output is 640x480 pixels (VGA) and 1280x720 pixels (HD). The camera has 70º visual angle with focus length of 4- 6cm and is water-resistant. The camera was taped to the Macintosh blade at a distance of 5 cm from the distal end of the blade, using transparent waterproof Leukofix® tape.
  Interventions: Device: Endotracheal intubation
- McGrath MAC® videolaryngoscope (McGrath) group (Active Comparator): The McGrath MAC® videolaryngoscope used in this study was equipped with disposable blade no.4
  Interventions: Device: Endotracheal intubation

INTERVENTIONS:
Device: Endotracheal intubation — Every eligible patient was intubated using either SAM-VL or McGrath MAC® according to their randomization allocation

SUMMARY:
Videolaryngoscopy highly improves success rate for endotracheal intubation in both normal and difficult airway. However, commercially available videolaryngoscope such as McGrath MAC® can be costly.

The. investigators aim to study a more economical alternative by comparing the intubation time, first attempt success rate, laryngeal visualization, complications, and user satisfaction between our self-assembled modified macintosh videolaryngoscope (SAM-VL) and McGrath MAC® (McGrath).

The study shows that endotracheal intubation using self-assembled modified videolaryngoscope is faster, had more successful first attempts, and allowed better glottis visualization compared with McGrath MAC®. It is a suitable alternative for videolaryngoscope in low resource setting.

DETAILED DESCRIPTION:
Background and Aims: Videolaryngoscopy highly improves success rate for endotracheal intubation in both normal and difficult airway. However, commercially available videolaryngoscope such as McGrath MAC® can be costly. The investigators aim to study a more economical alternative by comparing the intubation time, first attempt success rate, laryngeal visualization, complications, and user satisfaction between our self-assembled modified macintosh videolaryngoscope (SAM-VL) and McGrath MAC® (McGrath).

Settings and Design: This was a single-blind randomized clinical trial with 62 adult subjects. The investigators exclude patients with difficult airway, cardiac disease, and neuromuscular disease. The results were calculated using the Statistical Package for Social Scientists (SPSS) 24 Results: Median total intubation time was 63 s (27 - 114 s) in SAM-VL group, compared with 74 s (40 - 133 s), (p = 0,032) in McGrath group. The rate of successful first attempt in SAM-VL group was slightly higher than McGrath group at 90,3% vs 87.1%. Glottic visualization was more satisfactory in SAM-VL group with 67.7% of subjects having score of 100 and 29% of subject having score of 75. Complications found in this study were tachycardia (12.9% SAM-VL group vs 29% in McGrath group) and minimal airway mucosal laceration (9.7% in SAM-VL vs 3.2% in McGrath group). SAM-VL users rate the device high in ease of blade insertion and manoeuvrability, providing good laryngeal visualisation, and overall satisfaction rating.

Conclusions: Endotracheal intubation using self-assembled modified videolaryngoscope is faster, had more successful first attempts, and allowed better glottis visualization compared with McGrath MAC®.

Key-words: endotracheal intubation, self-assembled videolaryngoscope, McGrath MAC®, intubation time, glottis visualization Key Messages: Endotracheal intubation using self-assembled modified videolaryngoscope is faster, had more successful first attempts, and allowed better glottis visualization compared with McGrath MAC®. It is a suitable alternative for videolaryngoscope in low resource setting.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (18-65 years old), American Society of Anesthesiologists (ASA) physical status of I - II, Body Mass Index (BMI) of 18 - 30 kg/m2, scheduled for elective surgical procedures under general anesthesia

Exclusion Criteria:

* ASA III or above, difficult airway, pregnancy, cardiac condition, neuromuscular disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Time needed for Intubation "A" | After endotracheal intubation completed
  The time needed for Intubation "A" recording began when the tip of the laryngoscope blade passed through the incisors until the operator was able to achieve best visualization of the glottis. Measured in seconds (s).
Time needed for Intubation "B" | After the endotracheal intubation completed
  The time needed for Intubation"B" recording began when the operator received visualization of the glottis and ended after the endotracheal tube tube was confirmed to enter the trachea. Measured in seconds (s).
Total time needed for intubation | After the endotracheal intubation completed
  The sum total of time needed for Intubation A+B. Measured in seconds (s).

SECONDARY OUTCOMES:
Successful first attempt | After the endotracheal intubation completed
  Measuring intubation's first attempt success rate between the two groups. Success rate defined in number (%).
Laryngeal visualization | After the endotracheal intubation completed
  Measuring laryngeal visualization using Percentage of Glottic Opening (POGO) score: 100,75, 50, 25, 0.
Complications | After the endotracheal intubation completed
  Documenting complications generated by each device. Complications recorded are: Hypertension, hypotension, tachycardia, bradycardia, mucosal laceration, and esophageal intubation. Incidence are presented in numbers (%).
Laryngoscope User Satisfaction | After the endotracheal intubation completed
  Documenting laryngoscope user satisfaction in terms of blade insertion (very easy, easy, reasonable, difficult), device maneuverability (very easy, easy, reasonable, difficult), glottic visualization (very good, good, enough, poor), and overall satisfaction rating (very good, good, enough, poor).

CONTACTS AND LOCATIONS:
Overall Officials: Besthadi Sukmono, MD, Principal Investigator — Indonesia University
Locations (1):
- University of Indonesia and Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol and Statistical Analysis Plan
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data is available from 1 month after publication until 10 years
Access Criteria: by access

REFERENCES:
- [Background] Griesdale DE, Bosma TL, Kurth T, Isac G, Chittock DR. Complications of endotracheal intubation in the critically ill. Intensive Care Med. 2008 Oct;34(10):1835-42. doi: 10.1007/s00134-008-1205-6. Epub 2008 Jul 5. PMID 18604519
- [Background] Rosenblatt WH, Sukhupragarn W. Airway management. In: Barash PG, editor. Barash Clinical Anesthesia, 7th ed. Philadelphia:Lippincott William & Wilkins. 2013;27:763-778.
- [Background] Shin M, Bai SJ, Lee KY, Oh E, Kim HJ. Comparing McGRATH(R) MAC, C-MAC(R), and Macintosh Laryngoscopes Operated by Medical Students: A Randomized, Crossover, Manikin Study. Biomed Res Int. 2016;2016:8943931. doi: 10.1155/2016/8943931. Epub 2016 Sep 15. PMID 27703983
- [Background] Liu ZJ, Yi J, Guo WJ, Ma C, Huang YG. Comparison of McGrath Series 3 and Macintosh Laryngoscopes for Tracheal Intubation in Patients With Normal Airway by Inexperienced Anesthetists: A Randomized Study. Medicine (Baltimore). 2016 Jan;95(2):e2514. doi: 10.1097/MD.0000000000002514. PMID 26765472
- [Background] Wallace CD, Foulds LT, McLeod GA, Younger RA, McGuire BE. A comparison of the ease of tracheal intubation using a McGrath MAC((R)) laryngoscope and a standard Macintosh laryngoscope. Anaesthesia. 2015 Nov;70(11):1281-5. doi: 10.1111/anae.13209. Epub 2015 Sep 4. PMID 26336853
- [Background] Normand KC, Vargas LA, Burnett T, Sridhar S, Cai C, Zhang X, et al. Use of the McGRATH TM MAC : To view or not to view ?
- [Background] Ng I, Hill AL, Williams DL, Lee K, Segal R. Randomized controlled trial comparing the McGrath videolaryngoscope with the C-MAC videolaryngoscope in intubating adult patients with potential difficult airways. Br J Anaesth. 2012 Sep;109(3):439-43. doi: 10.1093/bja/aes145. Epub 2012 Jun 7. PMID 22677878
- [Background] Thong S, Teoh WH. Videolaryngoscopy and Indirect Intubating Aids in Airway Management. In: Khan Z, editor. Airway Management. 1st ed. Springer International Publishing Switzerland; 2014. p. 25-63
- [Background] Tanoubi I, Drolet P, Donati F. Optimizing preoxygenation in adults. Can J Anaesth. 2009 Jun;56(6):449-66. doi: 10.1007/s12630-009-9084-z. Epub 2009 Apr 28. PMID 19399574
- [Background] Karippacheril JG, Umesh G, Ramkumar V. Inexpensive video-laryngoscopy guided intubation using a personal computer: initial experience of a novel technique. J Clin Monit Comput. 2014 Jun;28(3):261-4. doi: 10.1007/s10877-013-9522-x. Epub 2013 Oct 17. PMID 24132806
- [Background] Latuconsina FW, Dedi Fitri Yadi S. Perbandingan intubasi endotrakea menggunakan clip-on smartphone camera videolaryngoscope dengan laringoskop Macintosh pada manekin. J Anestesi Perioper [Internet]. 2018;6(1):27-33
- See also: Xue FS, Li HX, Liu YY, Yang GZ. Current evidence for the use of C-MAC videolaryngoscope in adult airway management: A review of the literature. Ther Clin Risk Manag [Internet]. 2017;13:831-41 — http://www.embase.com/search/results?subaction=viewrecord&from=export&id=L617240527%0Ahttp://dx.doi.org/10.2147/TCRM.S136221
- See also: Walker L, Brampton W, Halai M, Hoy C, Lee E, Scott I, et al. Randomized controlled trial of intubation with the McGrath w Series 5 videolaryngoscope by inexperienced anaesthetists. Br J Anaesth [Internet]. 2009;103(3):440-5. — http://dx.doi.org/10.1093/bja/aep191
- See also: Levitan RM, Heitz JW, Sweeney M, Cooper RM. The Complexities of Tracheal Intubation With Direct Laryngoscopy and Alternative Intubation Devices. YMEM [Internet]. 2011;57(3):240-7. — http://dx.doi.org/10.1016/j.annemergmed.2010.05.035
- See also: Luqmanmuhamed M, Devadas P. Comparison between custom made video laryngoscope and Macintosh laryngoscope aided endotracheal intubation : a simple and inexpensive digital tool. IOSR J Dent Med Sci [Internet]. 2017;16(9):45-51. — http://www.iosrjournals.org
- See also: Hoshijima H, Mihara T, Maruyama K, Denawa Y, Takahashi M, Shiga T, et al. McGrath videolaryngoscope versus Macintosh laryngoscope for tracheal intubation: A systematic review and meta-analysis with trial sequential analysis. J Clin Anesth [Internet]. — http://doi.org/10.1016/j.jclinane.2017.12.030

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT04850976/Prot_SAP_ICF_000.pdf